CLINICAL TRIAL: NCT03577249
Title: Biological Effects of Citrate-buffered Solutions on Dialysis Efficiency and Systemic Inflammation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Vincenzo Cantaluppi, Associate professor of Nephrology, A.O.U. Città della Salute e della Scienza
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0064476; 2CEI-753 (Other: IRB from AO Citta Della Salute e Della Scienza di Torino)
Record Dates: First submitted 2018-06-13; First posted 2018-07-05 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Renal Insufficiency, Chronic; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation | interventions — Dialysis Solutions

STUDY DESIGN:
Intervention Model Description: 45 patients with end stage renal disease will be treated with dialysis solution A (standard of care: acetate-buffered) for 3 months then with solution B (acetate-free, citrate buffered, otherwise identical to solution A) for 3 months and then with solution A for the final 3 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Dialysis Solutions

INTERVENTIONS:
Drug: Dialysis Solutions — Solution A: 3mmol/L of acetate anion; Solution B: 1mmol/L of citrate anion

SUMMARY:
In this study 45 patients undergoing weekly dialysis for chronic end stage renal disease will be enrolled. The patients will be treated with a standard dialysis solution, containing acetate buffer, for 3 months; subsequently the acetate will be substituted with citrate anion for the 3 following months and then, the last 3 months, the standard acetate-solution will be restarted. The aim of the study is to assess if acetate-to-citrate switch in the dialysis solution influences dialysis efficiency and patient inflammatory state.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* creatinine clearance <5ml/min
* treatment with bicarbonate HD (BIC-HD) or on-line hemodiafiltration (OL-HDF) 3 times per week for at least 6 months prior to study start
* treated at Dialysis unit of: Città della Salute e della Scienza University Hospital, Torino, Italy

Exclusion Criteria:

* known neoplastic disease
* active chronic inflammatory disease
* active acute inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Change in serum CRP (C-reactive protein) | Months 4th to 6th
  Change in serum CRP during the 3 months of citrate-buffered dialysis

SECONDARY OUTCOMES:
Change in dialysis efficiency | Every 3 months (month 0, 6, 3 and completion - 9)
  Dougirdas formula will be used to estimate dialysis efficiency at the beginning and completion of each study interval
Change in serum CRP (C-reactive protein) | Every 3 months (month 0, 6, 3 and completion - 9)
  Variation of serum CRP at the beginning and completion of each study interval

CONTACTS AND LOCATIONS:
Locations (1):
- Città della Salute e Della Scienza di Torino - Presidi CTO e Molinette, Torino, To, Italy

IPD SHARING:
Plan to Share IPD: No